CLINICAL TRIAL: NCT05071989
Title: The Influence of Sleep Education Supported and Unsupported With Social Media Reminders on the Sleep Quality in Adolescents Aged 14-18: Randomized Controlled Study
Brief Title: The Influence of Sleep Education With Social Media Reminders on the Sleep Quality in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BAIBU-SBF-SC-01
Record Dates: First submitted 2021-09-15; First posted 2021-10-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Adolescent Behavior
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sleep education group do not supported with social media reminders (Experimental): Sleep education do not supported with social media reminders
  Interventions: Behavioral: Sleep Education
- Sleep education group supported with social media reminders (Experimental): Sleep education group supported with social media reminders
  Interventions: Behavioral: Sleep Education
- Control group (No Intervention): No intervention was made in the control group.

INTERVENTIONS:
Behavioral: Sleep Education — A single-blind school- based randomized controlled design
  Arms: Sleep education group do not supported with social media reminders; Sleep education group supported with social media reminders

SUMMARY:
Objective: This study aimed to determine the effect of sleep education, supported and unsupported with social media reminders, on sleep quality in 14-18 age group adolescents.

Design: This study is in a single-blind randomized controlled design. The study was carried out between October 2019 and January 2020.

Participants: The sample of this study consisted of 60 students randomly selected from three Anatolian High Schools in the city center. The students were divided into 3 groups of 20 people each (Experiment 1, Experiment 2, and Control). According to the scan result, adolescents who have sleep quality (PSQI>5 and CASQ>16), use Smartphone and the internet, have no chronic diseases and obesity, and have no mental problems were included in the study. Adolescents who use sleeping pills or any other medication and have communication obstacles were excluded from the study. The study was completed with 55 adolescents due to the separation of 5 adolescents during the experiment.

Intervention: The sleep education group, which was unsupported with social media reminders, was given sleep education for 30 minutes once a week for four weeks at school. In addition to the education at school, information messages and warnings were sent to the sleep education group, which was supported with social media reminders, via WhatsApp. The control group did not receive any intervention other than taking measurements of sleep parameters once a week.

Main Outcome(s) and Measure(s): The data were collected with Pittsburgh Sleep Quality Index, Cleveland Adolescent Sleepiness Questionnaire, Adolescent Sleep Habits Form and MI Band 3 device.

DETAILED DESCRIPTION:
The application of the research was planned according to the literature review and recommendations of the cognitive behavioral therapy approach. Sleep-related CBT practices consist of stimulus control, sleep restriction, relaxation techniques, managing sleep-related concerns, sleep hygiene education, and paradoxical intention. CBT practices consist of stimulus control and sleep hygiene education were used in this study. The sleep hygiene education that is part of the CBT method was used in the sleep education given to the Experiment 1 group. The sleep hygiene education that is part of the CBT method and the written stimulus control applications with WhatsApp was performed twice a day in the Experiment 2 group.

ELIGIBILITY:
Inclusion Criteria:

* Don't have any language and hearing problems
* Use the internet and Smartphone
* Do not have any chronic diseases
* Mental disorders and obesity
* Do not use any medication that causes sleep problems

Exclusion Criteria:

* Use sleeping pills
* Have psychiatric and chronic diseases
* Have mental disabilities were excluded from the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Sleep Quality | 4 weeks
  Pittsburgh Sleep Quality Index (PSQI):It is the most widely used scale to measure subjective sleep quality in the international literature. The scale was developed by Buyyse et al., in 1989, and validity and reliability studies in Turkish were carried out by Ağargün et al. The index has a diagnostic sensitivity of 89.6% and a specificity of 86.5%. The scale consists of a total of 18 items that make up 7 components. The maximum score that can be taken from the scale is 21. A score above 5 indicates poor sleep quality, while below 5 indicates good sleep quality.
Sleepiness | 4 weeks
  Cleveland Adolescent Sleepiness Questionnaire (CASQ): This scale provides a valid and reliable subjective measure that was used to determine the daytime sleepiness of adolescents aged 11-17 years. The scale was developed by Spilsbury et al., consists of 16 item questions measuring daytime sleepiness in adolescents. Scores range from 16 to 80 on a 5-point Likert-type scale (never: 1; rarely: 2; sometimes: 3; usually: 4; almost everyday: 5). Five of the statements are scored in the opposite direction. Daytime sleepiness is obtained by summing the scores of 16 items and the higher the score, the higher the daytime sleepiness. The high internal consistency of the scale (Cronbach's Alpha= 0.89) can be used both in clinical (for instance, in those with obstructive sleep apnea or OSA) and clinically healthy normal adolescents. The Turkish validity-reliability study of the scale was carried out in 2020 by Çağlar and Tokur Kesgin.
Sleep hygiene | 4 weeks
  Adolescent Sleep Habits Form (ASHF): According to the information obtained through the literature review, ASHF for sleep hygiene consisting of 33 questions for the adolescent age group was created. Opposite each question, some answers include "Never (0), rarely (1), Sometimes (2), Often (3) and Always (4)". The minimum score that can be taken from the questionnaire is 0, and the maximum is 132. It is conceivable that the higher the questionnaire score, the better the adolescent performs sleep hygiene practices. Davis' technique was used for the content validity of the questionnaire. To evaluate the survey questions in terms of scope, the opinions of 5 experts were consulted ( one of them is an assessment and evaluation specialist in education, four of them are faculty members from the field of nursing).
Sleep parameters | 4 weeks
  Xiaomi Mi Band 3 Sleeping Wristband: In the study, the sleep parameters of the students were followed by the Xiaomi Mi Band 3 actigraph wristband. Previous studies have proven that a wristband is a reliable device for measuring sleep parameters. This wristband was used as an actigraph for reasons such as a charging time of about two weeks, being waterproof, being compatible with Android devices and not requiring separate software for transferring data to a computer. The data on sleep parameters (total sleep time, deep and light sleep levels, time of falling asleep and waking up, time of sleep interruption) obtained in the study were recorded by the researcher every week from the students.

CONTACTS AND LOCATIONS:
Overall Officials: Songül Çağlar, PhD, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caglar S, Kesgin MT. The influence of sleep education supported and unsupported with social media reminders on the sleep quality in adolescents aged 14-18: a three-center, parallel-arm, randomized controlled study. Sleep Breath. 2024 Dec;28(6):2581-2590. doi: 10.1007/s11325-024-03138-6. Epub 2024 Sep 25. PMID 39320594